CLINICAL TRIAL: NCT00349778
Title: High-Dose Sequential Therapy and Single Autologous Transplantation for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sally Arai, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-05704; 97115 (Other: Stanford University Alternate IRB Approval Number); BMT183 (Other: OnCore number)
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Etoposide; etoposide phosphate; Melphalan; Carmustine; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- High-Dose Sequential Therapy (Experimental): Cyclophosphamide + Etoposide + Melphalan + Carmustine with Filgrastim
  Interventions: Drug: Cyclophosphamide; Drug: Etoposide; Drug: Melphalan; Drug: Carmustine; Drug: Filgrastim

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide as a white powder in 100 mg, 200 mg and 500 mg vials, to be dissolved in ~250 mL of saline or D5W and infused IV over 2 hours
  Other Names: Cytoxan; Neosar
Drug: Etoposide — 100 mg etoposide as 5 mL solution in clear ampules for injection.
  Other Names: Etopophos; VePesid; Toposar; VP-16; Etoposide phosphate
Drug: Melphalan — Melphalan as single-use glass vials of freeze-dried melphalan hydrochloride (equivalent to 50 mg of melphalan), to be reconstituted in 0.9% sodium chloride solution to not greater than 0.45 mg/mL, and administered within 1 hour of constitution.
  Other Names: Alkeran; L-PAM; L-Sarcolysin; Phenylalanine mustard
Drug: Carmustine — Carmustine as a powder for reconstitution in 100 mg vials, to be reconstituted with 3 mL sterile dehydrated ethanol and D5W. Carmustine should be dissolved in 500 mL of 5% dextrose in water (D5W) and infused IV over 2 hours.
  Other Names: BiCNU; BCNU
Drug: Filgrastim — Filgrastim in vials of 300 µg or 480 µg at a concentration of 300 µg/mL, to be given as a daily subcutaneous injection.
  Other Names: Neupogen; Granulocyte-colony stimulating factor (G-CSF)

SUMMARY:
This study uses a sequence of high-dose chemotherapy drugs and a stem cell transplant to treat multiple myeloma. The study is being performed to evaluate the efficacy and side effects of treatment. Specifically, the study is designed to reduce the risk of interstitial pneumonitis.

DETAILED DESCRIPTION:
Analysis of 196 previously treated patients demonstrated a median event-free survival (EFS) of 36 months with a median overall survival of more than 6 years. The main toxicity of this therapy is related to carmustine-induced pneumonitis or interstitial pneumonitis (IP). This complication is related to the dose of carmustine. Institutional experience in myeloma patients using this dose of carmustine indicates an incidence of IP of34%.

There have been recent studies evaluating the role of tandem autologous transplants for patients with multiple myeloma. These trials were based upon the hypothesis that performing tandem high-dose therapy regimens would lead to increased tumor cell kill, decreased tumor burden and an improvement in overall survival. Our results with high-dose sequential therapy including the dose-intense carmustine/melphalan transplant demonstrates similar median EFS and overall survival (OS) when compared with the results of tandem transplant approaches.The proposed trial will continue to use a high-dose sequential transplant approach, however, we will use a reduced dose of carmustine which we expect to be associated with a lower incidence of IP.

ELIGIBILITY:
INCLUSION CRITERIA

* Stage II to III multiple myeloma, or progression after initial treatment of Stage I disease; early or relapsed
* Age 18 to 75 years.
* Pathology reviewed and the diagnosis confirmed at Stanford University Medical Center.
* Patients with amyloidosis may be eligible for this trial, with approval by the Principle Investigator.
* Patients must have a Karnofsky performance status > 70%.
* Aspartate aminotransferase (AST) must be < 2 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) must be < 2 x ULN
* Total bilirubin < 2 mg/dL.
* Serum creatinine < 2.0 or 24-hour creatinine clearance ≥ 60 mL/min.
* Patients must be HIV-negative.
* Patients must provide signed, informed consent.

EXCLUSION CRITERIA

* Severe psychological or medical illness
* Prior autologous hematopoietic cell transplantation
* Pregnant
* Lactating women
* Smoldering multiple myeloma,
* Monoclonal gammopathy of unknown significance or primary amyloidosis will be excluded from this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-08; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally Arai, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen AI, Negrin RS, McMillan A, Shizuru JA, Johnston LJ, Lowsky R, Miklos DB, Arai S, Weng WK, Laport GG, Stockerl-Goldstein K. Tandem chemo-mobilization followed by high-dose melphalan and carmustine with single autologous hematopoietic cell transplantation for multiple myeloma. Bone Marrow Transplant. 2012 Apr;47(4):516-21. doi: 10.1038/bmt.2011.106. Epub 2011 May 23. PMID 21602899

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Dose Sequential Therapy
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all patients who proceeded to transplant on trial
Arm/Group | High-Dose Sequential Therapy
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 91
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 10
  Ethnicity: Not Hispanic or Latino | 85
  Ethnicity: Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pulmonary Toxicity
Description: Pulmonary toxicity was assessed as the incidence of interstitial pneumonitis.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Sequential Therapy
Number analyzed (Participants) | 102
Participants | 32

2. Secondary Outcome: Overall Participant Survival (OS)
Description: Survival status was assessed 5 years after transplant.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Sequential Therapy
Number analyzed (Participants) | 102
Participants | 52

3. Secondary Outcome: Number of Participants That Relapse After Autologous Transplantation
Description: Relapse was measured as the number of patients who relapse after high-dose sequential therapy then autologous transplantation
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | High-Dose Sequential Therapy
Number analyzed (Participants) | 102
Participants | 66

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | High-Dose Sequential Therapy
All-Cause Mortality (participants affected / at risk) | 22/102
Serious Adverse Events (participants affected / at risk) | 5/102
Other Adverse Events (participants affected / at risk) | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Sequential Therapy (N=102)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
aspergillus infection (Infections and infestations) | 1 (1)
Interstitial pneumonitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No